CLINICAL TRIAL: NCT04964817
Title: Heart Failure With Preserved Ejection Fraction (HFpEF) and Symptomatic Obstructive Iliofemoral Venous Disease and Venous Stenting: A Pilot Cohort Study
Brief Title: HFpEF and Symptomatic Obstructive Iliofemoral Venous Disease Study
Acronym: PERSUADE
Status: Terminated | Type: Observational
Why Stopped: unable to recruit following changes to practice resulting from pandemic
Sponsor: Prairie Education and Research Cooperative (Industry)
Collaborators: Boston Scientific Corporation (Industry); Medtronic (Industry); Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 1309580
Record Dates: First submitted 2021-06-18; First posted 2021-07-16 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Venous Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To ascertain the potential symptom improvement assessed by Cardiopulmonary Exercise Testing (CPET) in subjects with heart failure with preserved ejection fraction (HFpEF) and nonthrombotic iliofemoral venous lesions and/or iliocaval obstruction defined by MR or CT venography AND CEAP Clinical Category ≥3 prior to venous stenting.

DETAILED DESCRIPTION:
Primary Objective:

Evaluate potential improvement in metrics of functional capacity assessed by Cardiopulmonary Exercise Testing performed before and after venous stenting of an ≥50% iliofemoral venous obstruction by MR or CT venography and confirmed by intra-procedural IVUS in a prospective patient cohort presenting with heart failure with preserved ejection fraction with a H2FpEF score of ≥4 AND a CEAP Category ≥3.

Secondary Objectives:

Identify patient demographic, baseline laboratory, imaging, procedural and Cardiopulmonary Exercise Testing variables and the FDA-approved Minnesota Living with Heart Failure Questionnaire as a Medical Device Development Tool (MDDT) in patients with and without functional improvement as assessed by Cardiopulmonary Exercise Testing VO2max after successful venous stenting of iliofemoral/iliocaval venous obstructions.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent and comply with all study requirements
* Age ≥ 40 years of age
* Stable, symptomatic heart failure with preserved ejection fraction and a H2FpEF Score ≥4
* Presence of non-malignant inferior vena cava obstruction, a unilateral or bilateral chronic non-malignant obstruction of the common femoral vein, external iliac vein, common iliac vein, or any combination thereof, defined as a ≥50% reduction in target vessel lumen diameter defined by screening MRV, CTV and confirmed by a 50% reduction in luminal area as assessed by intraprocedural IVUS.
* Previous (>6 months) history of ilio-femoral and/or lower extremity deep venous thrombosis associated with a residual ilio-femoral venous obstruction ≥50% by MRV, CTV.
* Clinically significant venous obstruction meeting CEAP Clinical classification ≥3.
* Negative pregnancy test in females of child-bearing potential

Exclusion Criteria:

* Subject hospitalized for acute compensated heart failure within 60 days prior to enrollment
* Presence of history of clinically significant pulmonary emboli within 6 months prior to enrollment.
* Subject has any permanent neurologic defect that may cause non-compliance with the protocol
* Subject has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematous).
* Subject has an allergy to contrast media that cannot be adequately pre-treated prior to the required diagnostic and/or endovascular procedures.
* Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding.
* Subject has renal failure or chronic kidney disease with glomerular filtration rate (GFR) ≤ 30 mL/min or Modification of Diet in Renal Disease (MDRD) study equation result of ≤ 30 mL/min per 1.73 m2.
* Subject has white blood cell (WBC) count < 3.0 (3000 cells/mm3) within 7 days prior to index procedure.
* Subject has a platelet count < 80,000 cells/mm3 or > 700,000 cells/mm3 ≤ 7 days pre procedure; uncorrected hemoglobin of ≤9 g/dL.
* Subject has known or suspected active systemic infection evidenced by WBC > 14.0 (14,000/mm3).
* Subject is currently participating in another investigational drug or device study.
* Subject intends to participate in another investigational drug or device study within 30 days after the index procedure.
* Subject has moderate or severe pulmonary disease (i.e., COPD) considered by Investigator to be a major contributing factor to the subject's exertional dyspnea

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients ≥40 years old with diagnosed HFpEF by established standard of care clinical ACC/AHA Congestive Heart Failure Definition and Clinical Guidelines23 and a Mayo Clinic H2FpEF Score ≥ 4 with evidence of peripheral venous disease assessed by the CEAP Classification 3 according to the Reporting Standards of International Society of Cardiovascular Surgery (ISCV)/Society of Vascular Society (SVS).24
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Evaluate potential change in metrics of functional capacity assessed by Cardiopulmonary Exercise Testing performed before and after venous stenting | 180 days
  The primary focus of the study is to estimate the change in functional capacity in patients of heart failure with preserved ejection fraction (HFpEF) of varying severities and chronic peripheral venous disease associated with pelvic venous obstruction after resolution via IVUS-guided venous stenting. Key estimate will be the change in functional capacity (i.e., VO2max or 6MWD) as assessed by the percentage change in pre- and post-venous stenting. No formal hypothesis tests are pre-specified.

SECONDARY OUTCOMES:
Identify patient functional change utilizing the FDA-approved Minnesota Living with Heart Failure Questionnaire as a Medical Device Development Tool (MDDT) post treatment versus pre treatment | 180 days
  The secondary outcome measure of the study is to estimate the change in functional capacity in patients of heart failure with preserved ejection fraction (HFpEF) of varying severities and chronic peripheral venous disease associated with pelvic venous obstruction after resolution via IVUS-guided venous stenting. Key estimate will be the change in functional capacity as assessed by the percentage change in pre- and post-venous stenting utilizing the Minnesota Living with Heart Failure Questionnaire (MLHFQ). No formal hypothesis tests are pre-specified.

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Rocha-Singh, MD, Principal Investigator — Prairie Cardiovascular Consultants
Locations (1):
- Prairie Heart Institute at St. Johns Hospital, Springfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No